CLINICAL TRIAL: NCT01996046
Title: 18F-fluorodeoxyglucose (FDG) Positron Emission Tomography (PET/CT) for the Evaluation of Response to Therapy in Bone-dominant Metastatic Breast Cancer
Brief Title: FDG PET/CT in Breast Cancer Bone Mets
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 817940; UPCC17113 (Other: Penn cancer center); NCT02110160 (obsolete NCT alias)
Record Dates: First submitted 2013-11-08; First posted 2013-11-27 (Estimated); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Estrogen Receptor Positive Breast Cancer; Bone Metastases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Bone mets: Patients will undergo an [18F] FDG PET/CT scan at 4 weeks after starting new hormonal therapy
  Interventions: Other: FDG PET/CT scan

INTERVENTIONS:
Other: FDG PET/CT scan — [18F] FDG PET/CT scan at 4 weeks after starting new hormonal therapy

SUMMARY:
This study will evaluate baseline uptake on a FDG PET/CT scan in patients with breast cancer that has spread to the bones. A repeat FDG PET/CT scan will be done 4 weeks after the start of new breast cancer hormone treatment and again at 12 weeks after treatment start. The baseline uptake and change in uptake after the repeat scans will be compared to clinical long term outcomes such as time to progression and overall survival. In addition the uptake will be compared to the incidence of skeletal related events that are common occurrences in patients with cancer that has spread to the bones.

DETAILED DESCRIPTION:
This is an observational study as all patients will receive the same research diagnostic test, an FDG PET/CT study performed at 4 weeks after starting new hormone treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients, at least 18 years of age, with a history of pathologically confirmed ER+ breast cancer
2. Biopsy proven or clinically obvious documented bone metastases from breast cancer (with the majority of the disease burden in the bone)
3. Patients planning to start new endocrine targeted therapy (any line of therapy is acceptable and any endocrine therapy is allowed)
4. Willing and able to comply with scheduled visits and serial imaging procedures
5. Agrees to allow access to clinical records regarding response to treatment and long term follow up.
6. Be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines

Exclusion Criteria:

1. Women who are pregnant or breast feeding
2. Uncontrolled diabetes mellitus (fasting glucose greater than 200 mg/dL)
3. Inability to tolerate imaging procedures (e.g. claustrophobia, severe pain)
4. Weight exceeding capacity of imaging table
5. Previous treatment with radiation or surgery to a significant percentage of bony metastatic sites
6. Treatment with marrow stimulating agents (e.g. granulocyte colony stimulating factor (GCSF)) within 3 weeks of baseline scan

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a history of ER+ breast cancer with documented bone metastases from breast cancer. Patients must be planning to start new hormone therapy for their breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2013-09; Primary Completion 2023-07-31 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | medical record reviewed every 6 months from date of enrollment to date of progression, up to 120 months
  Date of clinical progression will be recorded

SECONDARY OUTCOMES:
Overall Survival | medical record reviewed every 6 months from date of enrollment to date of death, up to 120 months
  Date of death will be recorded

OTHER OUTCOMES:
Number of patients who have a Skeletal Related Event | medical record reviewed every 6 months from date of enrollment to date of death, up to 120 months
  Occurrence of radiation therapy to stabilize skeletal disease, pathologic fracture,spinal cord compression, surgery to stabilize the skeleton or hypercalcemia of malignancy will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: David Mankoff, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Hospital, Philadelphia, Pennsylvania, United States